CLINICAL TRIAL: NCT02696668
Title: The Effect of a Modified FaME vs. a Multisensory Group Balance Programme on Falls Risk, Balance Confidence and Quality of Life in Older Adult Who Fall or Are at Risk of Falling
Brief Title: Advances in Group-based Falls Rehabilitation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: King's College London (Other)
Collaborators: University College London Hospitals (Other); Guy's and St Thomas' NHS Foundation Trust (Other); St George's University Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KingsCL
Record Dates: First submitted 2016-02-25; First posted 2016-03-02 (Estimated); Last update posted 2017-03-10 (Actual); Status verified 2017-03

CONDITIONS: Accidental Falls
Keywords: multisensory exercises; group-based balance exercise programme

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- modified FaME (Active Comparator): Participants in the modified FaME group will receive a 16 weeks falls rehabilitation programme which will be tailored and progressed according to their abilities and their needs by the physiotherapist / instructor providing the rehabilitation at the hospital.
  Interventions: Other: modified FaME
- Multisensory (Experimental): Participants in the multisensory group will receive balance exercises training which will be tailored and progressed to their abilities and needs.
  Interventions: Other: Multisensory

INTERVENTIONS:
Other: modified FaME — Group based exercise classes one hour weekly for 16 weeks. Each exercise class will have 8-10 participants and two instructors. The components of the FaME programme include specific falls management strategies, such as bone loading, gait, dynamic posture, balance, reaction and co-ordination training, functional floor activities to improve coping skills and confidence.
  Arms: modified FaME
Other: Multisensory — Group based exercise classes one hour weekly for 16 weeks. Each exercise class will have 8-10 participants and two instructors.Participants will receive an initial assessment by the research physiotherapists to determine the most appropriate interventions for each participant. Interventions used will include:
  1. Limits of stability training with eyes open / eyes closed
  2. Self induced movement strategies with eyes open / eyes closed
  3. Gaze stability exercises in sitting / standing / walking
  4. Sensory integration
  5. Habituation exercises
  Arms: Multisensory

SUMMARY:
This study's main aim is to compare the effect of a modified FaME vs. a multisensory balance exercise programme on falls risk, balance confidence and quality of life in older adults who fall or at risk of falling when implemented in a group setting.

DETAILED DESCRIPTION:
Falls in older adults have a major impact on health, morbidity and mortality and have significant cost implications to healthcare providers (Alexander et al., 1992, Tinetti and Williams, 1998, Davis et al., 2010). Government legislation states targeted multifactorial falls rehabilitation programmes should be provided to older adult fallers (Excellence, 2013). The FaME programme, a group based rehabilitation programme is reported effective for improving balance and walking speed, and reducing the number of falls, chance of hospitalization, institutionalization, and death, and fear of falling (Skelton et al., 2005, Yeung et al., 2014). Sensory integration and re-weighting of peripheral sensory information from visual, somatosensory, and vestibular (i.e. inner ear) systems play an important role in maintaining balance (Horak, 2006). However, until recently no studies had incorporated vestibular exercises into falls rehabilitation programmes and therefore, the efficacy of this type of multisensory balance programme in older adult fallers was unknown.

A recent study showed that a programme combining the widely used modified OTAGO falls rehabilitation programme with multisensory balance exercises was feasible in older adult fallers and may have a greater beneficial effect on balance, gait, and falls risk compared to the OTAGO programme in isolation (Liston et al., 2014). However, multisensory rehabilitation targeting sensory integration and re-weighting which is crucial for postural control is not addressed in current guidelines. To develop the best programme for fall prevention, understanding the complexity of postural control and defining a specified exercise programme targeting essential systems is required. The FaME programme includes certain multisensory balance exercises, but these are introduced only in the latter phase of the programme. This study's main aim is to compare the effect of a modified FaME vs. a multisensory balance exercise programme on falls risk, balance confidence and quality of life in older adults who fall or at risk of falling when implemented in a group setting.

Research questions:

Primary research question:

Does exposure to multisensory balance rehabilitation provide better outcome in balance confidence, falls risk and quality of life in older adult who fall or are at risk of falling compared to the modified FaME programme?

Secondary research questions:

1. What is the long term effect of a multisensory balance rehabilitation programme vs. the modified FaME on all outcome measure scores and falls rate?
2. Is there a relationship between baseline cognitive function, vestibular function and intervention outcome?
3. Can vestibular dysfunction be effectively screened for in a community setting?

Study design:

This study will be a single blinded randomised control study to investigate the effect of the multisensory balance rehabilitation programme vs. the modified FaME on falls risk, balance confidence and quality of life in older adults who fall or are at risk of falling. This study will have two arms provided within a community-based setting. This study will compare intervention outcome between participants receiving the modified FaME falls rehabilitation programme and those receiving multisensory balance rehabilitation exercises.

ELIGIBILITY:
Inclusion Criteria:

Older adult 65 years old or older who have either experienced a fall or are at risk of falling (Timed Up and Go score >15 seconds) and have been referred by the assessing physiotherapist to a falls rehabilitation group class.

Exclusion Criteria:

1. Older adults who have:

   i) Cardiac syncope/pre-syncope ii) Postural hypotension iii) A Mini Mental State score of <24/30. ii) Diagnosis of dementia or mild cognitive impairment ii) Acute illness iii) Side effects of medication or drug intoxication iv) Evident musculo-skeletal or neurological deficit that is likely to contribute to postural instability
2. Any individual with poor written/spoken English will not be included in the study due to the need to complete multiple questionnaires.
3. Individuals with a known history of epilepsy in the last one year or currently experiencing migraine will not be included in this study due to the use of optokinetic stimuli.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-05-01 (Estimated); Primary Completion 2019-12-01 (Estimated); Study Completion 2020-03-01 (Estimated)

PRIMARY OUTCOMES:
Functional Gait Assessment | Baseline (prior to start of intervention), 8 weeks, 16 weeks and 32 weeks
  A 10-item test assesses complex gait tasks such as walking with head turns or stepping over an obstacle

SECONDARY OUTCOMES:
Timed Up and Go test | Baseline (prior to start of intervention), 8 weeks, 16 weeks and 32 weeks
  A validated test of balance used to examine functional mobility.
Mini Balance Evaluation Systems Test | Baseline (prior to start of intervention), 8 weeks, 16 weeks and 32 weeks
  A validated test designed to assess multiple aspects of postural control systems that may contribute to poor functional balance in adults
Activities-Specific Balance Confidence Scale | Baseline (prior to start of intervention), 8 weeks, 16 weeks and 32 weeks
  A validated self-report scale to assess balance confidence in daily activities
Falls Efficacy Scale - International | Baseline (prior to start of intervention), 8 weeks, 16 weeks and 32 weeks
  A validated self-report measure of fear of falling that assesses both easy and difficult physical and social activities
Environmental Analysis of Mobility Questionnaire | Baseline (prior to start of intervention), 8 weeks, 16 weeks, 32 weeks and one year
  A validated self-report scale to assess the relationship between characteristics of the physical environment and mobility disability
Hospital Anxiety and Depression Scale | Baseline (prior to start of intervention), 8 weeks, 16 weeks, 32 weeks and one year
  A self-report scale to assess anxiety and depression symptom.
EQ-5D self-report questionnaire | Baseline (prior to start of intervention), 8 weeks, 16 weeks, 32 weeks and one year
  A standardised measure of health outcome.
Vestibular Symptom Scale | Baseline (prior to start of intervention), 8 weeks, 16 weeks, 32 weeks and one year
  A validated self-report scale to assess common vestibular symptoms (i.e. giddiness) and autonomic/somatic anxiety symptoms.

OTHER OUTCOMES:
Cantab Dementia Battery | Baseline (prior to start of intervention), 8 weeks, 16 weeks and 32 weeks
  A validated computerized cognitive assessment system for measuring the severity of cognitive impairment in patients with prodromal Alzheimer's disease and those functioning within the dementia range

CONTACTS AND LOCATIONS:
Overall Officials: Marousa Pavlou, PhD, Principal Investigator — King's College London

IPD SHARING:
Plan to Share IPD: Undecided